CLINICAL TRIAL: NCT03105167
Title: Transforaminal Lumbar Interbody Fusion With Cortical Bone Trajectory Screws vs. Traditional Pedicle Screws Fixation: a Multicentre Randomised Controlled Trial
Brief Title: Cortical Bone Trajectory Screws vs. Traditional Pedicle Screws Fixation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Wenfei Ni, director, Second Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2017-08-106
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Spinal Stenosis Lumbar; Lumbar Disc Herniation; Intervertebral Disc Degeneration
Keywords: CBT; RCT; TLIF
MeSH Terms: conditions — Intervertebral Disc Displacement; Intervertebral Disc Degeneration | interventions — Pedicle Screws

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-TLIF group (Experimental): Patients who are randomised to the CBT-TLIF group will have cortical bone trajectory screws instead of pedicle screws During the opreation. After preventive use of antibliotics,A small skin incision was made at the fused segment, an entry point for insertion of the CBT screws was drilled in the junction of the center of the superior articular process and 1 mm inferior to the inferior border of the transverse process according to Matsukawa et al.A straight probe was used to create a trajectory for the CBT screws from the entry point to the opposite corner of the pedicle and vertebral body under anteroposterior fluoroscopic guidance.nilateral facetectomy is performed to gain access to the intervertebral disc.Afterwards, interbody fusion was performed.Device: CBT screws.
  Interventions: Procedure: cortical bone trajectory screws
- PS-TLIF group (Experimental): Patients who are randomised to the PS-TLIF group will have pedicle screws During the opreation. A posterior midline incision, about 6 cm, was performed at the level of interest level under fluoroscopic guidance. Pedicle screws were inserted into the vertebral body by using freehand, and the inferior and superior articular processes and part pf the lamina were removed by using an osteotome. To expose the lateral border of the ipsilateral nerve root, the ligamentum flavum was removed. Afterwards, interbody fusion was performed.Device:traditional pedicle screws.
  Interventions: Procedure: pedicle screws

INTERVENTIONS:
Procedure: cortical bone trajectory screws — cortical bone trajectory screws fixation takes the place of traditional pedicle screws fixation will be used in transforaminal lumbar interbody fusion.
  Arms: CBT-TLIF group
Procedure: pedicle screws — traditional pedicle screws fixation will be used in transforaminal lumbar interbody fusion.
  Arms: PS-TLIF group

SUMMARY:
Transforaminal lumbar interbody fusion (TLIF) had been favorable for effectively decrease pain and disability in specific spinal disorders; however, there has been concern regarding pedicle screw placement during TLIF surgery. Recently, several biomechanical studies had demonstrated that CBT technique achieves screw purchase and strength equivalent to or greater than the traditional method. Furthermore, Only 1 report examined the surgical outcomes of TLIF with CBT screws fixation compared with TLIF using traditional pedicle screws fixation. TLIF with CBT screws fixation may be effective for specific spinal disorders, but the evidence supporting this possibility is still limited.

DETAILED DESCRIPTION:
Methods and analysis: Blinded Randomized Controlled Trial (RCT) will be conducted. A total of 108 participants will be randomly allocated to either a CBT-TLIF group or a PS-TLIF group at a ratio of 1:1. The primary clinical outcome measures are: change in back and lower limb pain with Visual analogue scale (VAS) and change in quality adjusted life years (QALY) will be assessed by EQ-5D-5L. Measurements will be carried out at five fixed time points (pre-operatively and at 3, 6, 12 and 24 months).

Ethics and dissemination: The study had been reviewed and approved by the ethics committee of the Second affiliated hospital of the Wenzhou Medical University, Wenzhou, China(batch:2017-03). The results will be presented in peer-reviewed journals and related website within 2 years after the last operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years;
2. All of participants will be informed consent;
3. Chronic low back pain (visual analogue scale at least 3 out of 10 at rest and at least 5 out of 10 under physical strain) after having failed conservative treatment for 6 months;
4. Single-segment lower lumbar vertebral disease (Including lumbar spinal cannal stenosis, foraminal stenosis, segmental instability, lumbar disc herniation, and painful disc degeneration (back disc);

Exclusion Criteria:

1. Serious deformity of lumbar vertebrae;
2. Dysplasia of lumbar pedicle or vertebral laminar;
3. Obvious osteoporosis of lumbar vertebrae;
4. Metabolic bone diseases such as osteomalacia or Paget's disease;
5. Spondylolisthesis > grade 2 (Meyerding);
6. Caudaequina injury or severe radiculopathy;
7. Post inflammatory instability of the vertebral spine;
8. Body mass index > 30;
9. Immunologic diseases or Metabolic syndrome;
10. Therapy with systemic corticosteroids or immunosuppressants;
11. Current using Coumadin (or Warfarin) or Heparin therapy for more than 6 months at the time of operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-12-13 (Estimated); Study Completion 2021-12-13 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale(VAS) | up to 36 months
  pain score

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | up to 48 months
  The Oswestry Disability Index pain score
Symptomatic adjacent-segment disease (SASD) | up to 48 months
  Symptomatic adjacent-segment disease rate
Japanese Orthopedic Association (JOA) | up to 48 months
  Japanese Orthopedic Association score

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
All of the patients' outcomes (without patients' personal information) will be public shared within 2 years after clinical trial complete.

REFERENCES:
- [Result] Resnick DK, Choudhri TF, Dailey AT, Groff MW, Khoo L, Matz PG, Mummaneni P, Watters WC 3rd, Wang J, Walters BC, Hadley MN; American Association of Neurological Surgeons/Congress of Neurological Surgeons. Guidelines for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 8: lumbar fusion for disc herniation and radiculopathy. J Neurosurg Spine. 2005 Jun;2(6):673-8. doi: 10.3171/spi.2005.2.6.0673. PMID 16028736
- [Result] Brayda-Bruno M, Tibiletti M, Ito K, Fairbank J, Galbusera F, Zerbi A, Roberts S, Wachtel E, Merkher Y, Sivan SS. Advances in the diagnosis of degenerated lumbar discs and their possible clinical application. Eur Spine J. 2014 Jun;23 Suppl 3:S315-23. doi: 10.1007/s00586-013-2960-9. Epub 2013 Aug 27. PMID 23978994
- [Result] Omidi-Kashani F, Hasankhani EG, Ashjazadeh A. Lumbar spinal stenosis: who should be fused? An updated review. Asian Spine J. 2014 Aug;8(4):521-30. doi: 10.4184/asj.2014.8.4.521. Epub 2014 Aug 19. PMID 25187873
- [Result] Harms JG, Jeszenszky D. Die posteriore, lumbale, interkorporelle Fusion in unilateraler transforaminaler Technik. Oper Orthop Traumatol. 1998 Jun;10(2):90-102. doi: 10.1007/s00064-006-0112-7. No abstract available. German. PMID 17332991
- [Result] Rouben D, Casnellie M, Ferguson M. Long-term durability of minimal invasive posterior transforaminal lumbar interbody fusion: a clinical and radiographic follow-up. J Spinal Disord Tech. 2011 Jul;24(5):288-96. doi: 10.1097/BSD.0b013e3181f9a60a. PMID 20975594
- [Result] Santoni BG, Hynes RA, McGilvray KC, Rodriguez-Canessa G, Lyons AS, Henson MA, Womack WJ, Puttlitz CM. Cortical bone trajectory for lumbar pedicle screws. Spine J. 2009 May;9(5):366-73. doi: 10.1016/j.spinee.2008.07.008. Epub 2008 Sep 14. PMID 18790684
- [Result] Matsukawa K, Yato Y, Kato T, Imabayashi H, Asazuma T, Nemoto K. In vivo analysis of insertional torque during pedicle screwing using cortical bone trajectory technique. Spine (Phila Pa 1976). 2014 Feb 15;39(4):E240-5. doi: 10.1097/BRS.0000000000000116. PMID 24253778
- [Result] Baluch DA, Patel AA, Lullo B, Havey RM, Voronov LI, Nguyen NL, Carandang G, Ghanayem AJ, Patwardhan AG. Effect of physiological loads on cortical and traditional pedicle screw fixation. Spine (Phila Pa 1976). 2014 Oct 15;39(22):E1297-302. doi: 10.1097/BRS.0000000000000553. PMID 25099320
- [Result] Perez-Orribo L, Kalb S, Reyes PM, Chang SW, Crawford NR. Biomechanics of lumbar cortical screw-rod fixation versus pedicle screw-rod fixation with and without interbody support. Spine (Phila Pa 1976). 2013 Apr 15;38(8):635-41. doi: 10.1097/BRS.0b013e318279a95e. PMID 23104197
- [Result] Matsukawa K, Kato T, Yato Y, Sasao H, Imabayashi H, Hosogane N, Asazuma T, Chiba K. Incidence and Risk Factors of Adjacent Cranial Facet Joint Violation Following Pedicle Screw Insertion Using Cortical Bone Trajectory Technique. Spine (Phila Pa 1976). 2016 Jul 15;41(14):E851-E856. doi: 10.1097/BRS.0000000000001459. PMID 26796712
- [Result] Kasukawa Y, Miyakoshi N, Hongo M, Ishikawa Y, Kudo D, Shimada Y. Short-Term Results of Transforaminal Lumbar Interbody Fusion Using Pedicle Screw with Cortical Bone Trajectory Compared with Conventional Trajectory. Asian Spine J. 2015 Jun;9(3):440-8. doi: 10.4184/asj.2015.9.3.440. Epub 2015 Jun 8. PMID 26097661
- [Result] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Result] Matsukawa K, Yato Y, Nemoto O, Imabayashi H, Asazuma T, Nemoto K. Morphometric measurement of cortical bone trajectory for lumbar pedicle screw insertion using computed tomography. J Spinal Disord Tech. 2013 Aug;26(6):E248-53. doi: 10.1097/BSD.0b013e318288ac39. PMID 23429319
- [Result] Dixon JS, Bird HA. Reproducibility along a 10 cm vertical visual analogue scale. Ann Rheum Dis. 1981 Feb;40(1):87-9. doi: 10.1136/ard.40.1.87. PMID 7469530
- [Result] M Versteegh M, M Vermeulen K, M A A Evers S, de Wit GA, Prenger R, A Stolk E. Dutch Tariff for the Five-Level Version of EQ-5D. Value Health. 2016 Jun;19(4):343-52. doi: 10.1016/j.jval.2016.01.003. Epub 2016 Mar 30. PMID 27325326
- [Result] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Result] Okuda S, Miyauchi A, Oda T, Haku T, Yamamoto T, Iwasaki M. Surgical complications of posterior lumbar interbody fusion with total facetectomy in 251 patients. J Neurosurg Spine. 2006 Apr;4(4):304-9. doi: 10.3171/spi.2006.4.4.304. PMID 16619677
- [Result] Hagg O, Fritzell P, Nordwall A; Swedish Lumbar Spine Study Group. The clinical importance of changes in outcome scores after treatment for chronic low back pain. Eur Spine J. 2003 Feb;12(1):12-20. doi: 10.1007/s00586-002-0464-0. Epub 2002 Oct 24. PMID 12592542
- [Result] Ostelo RW, de Vet HC. Clinically important outcomes in low back pain. Best Pract Res Clin Rheumatol. 2005 Aug;19(4):593-607. doi: 10.1016/j.berh.2005.03.003. PMID 15949778
- [Derived] Wu C, Hu X, Liu R, Xu C, Jiang Y, Ge Z, Zhou K, Zhang D, Wu A, Dou H, Xu H, Tian N, Hu Z, Ni W. Comparison of the clinical and radiographic outcomes of cortical bone trajectory and traditional trajectory pedicle screw fixation in transforaminal lumbar interbody fusion: a randomized controlled trial. Eur Spine J. 2024 Mar;33(3):1069-1080. doi: 10.1007/s00586-023-08086-5. Epub 2024 Jan 22. PMID 38246903
- [Derived] Feng Z, Li X, Tang Q, Wang C, Zheng W, Zhang H, Wu AM, Tian N, Wu Y, Ni W. Transforaminal lumbar interbody fusion with cortical bone trajectory screws versus traditional pedicle screws fixation: a study protocol of randomised controlled trial. BMJ Open. 2017 Oct 22;7(10):e017227. doi: 10.1136/bmjopen-2017-017227. PMID 29061616